CLINICAL TRIAL: NCT04729920
Title: Predictors of Home Use of Mechanical Insufflation/Exsufflation Devices in Neuromuscular Patients: a Cross-sectional Study
Brief Title: Home Use of Mechanical Insufflation/Exsufflation Devices in Neuromuscular Diseases
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Ligue Pulmonaire Vaudoise (Unknown); University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, GEORGIA MITROPOULOU, Cheffe de clinique, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2019-01114
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Neuromuscular Diseases
Keywords: Mechanical insufflation-exsufflation; Cough assistance
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- subjects with neuromuscular disease: Adult subjects with neuromuscular disease, with an active prescription of MI-E for more than 3 months
  Interventions: Device: Mechanical insufflation/exsufflation device (MI-E)

INTERVENTIONS:
Device: Mechanical insufflation/exsufflation device (MI-E) — download of device (MI-E) data and self-reported satisfaction with the device

SUMMARY:
With this cross-sectional study of adult subjects with neuromuscular disease in the French-speaking part of Switzerland, we aim to explore MI-E adherence using self-report questionnaires and device data in order to identify the factors that influence the pattern of MI-E use and satisfaction with the treatment. Determining potential barriers to regular long-term home use of MI-E could help in identifying the patients who would benefit most from this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Diagnosis of neuromuscular disease
* Active prescription of MI-E for more than 3 months

Exclusion Criteria:

-Invasive airway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with neuromuscular disease, with an active prescription of MI-E for more than 3 months
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Adherence to MI-E (reported) | 12 months, or since treatment initiation (> 3 months)
  based on self-reported use
Adherence to MI-E (objective) | 12 months, or since treatment initiation (> 3 months)
  based on data downloads

SECONDARY OUTCOMES:
Satisfaction with the device | 12 months, or since treatment initiation (> 3 months)
  Self-report questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie, CHUV, Lausanne, Canton of Vaud, Switzerland